CLINICAL TRIAL: NCT01673802
Title: The Role of Gadoxetate Enhanced Spectral Dual-Energy CT in Evaluating Hilar Cholangiocarcinoma
Brief Title: The Role of Gadoxetate (Eovist) Enhanced CT in Evaluating Cholangiocarcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Society of Abdominal Radiology (Other)
Responsible Party: Principal Investigator, John V. Thomas, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R11-153; 117354 (Other: FDA)
Record Dates: First submitted 2012-08-13; First posted 2012-08-28 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Single arm study, with dose adjustment.
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT imaging (Experimental): Patients will undergo a standard of care Gadoxetate (Eovist) MRI for cholangiocarcinoma. Patients will then be immediately placed on the CT scanner. Patients will undergo a dual energy CT of the abdomen with no additional contrast.
  Interventions: Drug: CT scan

INTERVENTIONS:
Drug: CT scan — Gadoxetate (Eovist) enhanced dual energy CT
  Other Names: Dual Energy CT

SUMMARY:
The purpose of this project is to evaluate the role of gadoxetate (Eovist®) enhanced dual-energy CT in better evaluating perihilar cholangiocarcinoma. This pilot project aims to address a long-term pitfall in the imaging of cholangiocarcinomas, by providing higher resolution delineation of these often infiltrative tumors on single-source, Dual-Energy Spectral Multi Detector CT (MDCT), capitalizing on improved spatial resolution achievable with MDCT compared to MRI and at the same time producing a non-invasive CT cholangiogram to aid in accurate diagnosis and treatment planning of cholangiocarcinoma, particularly, the hilar variety.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the role of gadoxetate (Eovist) enhanced dual-energy CT in better evaluating perihilar cholangiocarcinoma, by exploiting the combination of the physiologic behavior of gadoxetate in liver tissue combined with the advantageous mass attenuation coefficient of Gadolinium achievable through dual energy technique. This combination of unique CT imaging sensitivity, high resolution and differential enhancement potentially allows improved visualization and detection of tumor relative to enhancing surrounding hepatic parenchyma and ductal anatomy in the hepatobiliary phase, due to the biliary excretion of the agent.

Cholangiocarcinoma is a hepatic adenocarcinoma that arises from the bile duct epithelium and is the second most prevalent liver cancer after hepatocellular carcinoma. The hilar intrahepatic variety of cholangiocarcinoma can present as an infiltrative, exophytic, or polypoid lesion. Most extra-hepatic cholangiocarcinomas are infiltrative, causing a focal stricture of the bile duct and result in proximal biliary ductal dilatation.

While magnetic resonance (MR) cholangiography is diagnostic in the majority of patients with malignant hilar strictures, evaluation is limited by spatial resolution and in some patients, the inability to have an MRI scan. Standard Multi Detector CT (MDCT) using iodinated contrast agents, on the other hand, is limited in evaluation of cholangiocarcinomas, due to the lack of consistent enhancement of the tumor with iodinated contrast.

Single-source, Dual-Energy (SSDE) Spectral MDCT utilizes a single fast switching x-ray beam source to acquire near simultaneous data sets at two different photon energies during a single acquisition. Data is acquired at 80 kilovolt peak (kVp) and 140 kVp with image reconstruction achievable as a selectable monochromatic presentation over a range of 40 - 140 kiloelectron volt (keV), typically 70-78 keV for diagnostic image presentation. At lower tube voltage, the frequency of photoelectric interactions increases exponentially and is strongly dependent on the atomic number. Therefore, for substances with higher atomic number, such as iodine and gadolinium the increased frequency of photoelectric and k-edge interactions at low tube voltage substantially increases CT attenuation, thus improving contrast. Gadolinium is further unique with k-edge attenuation at approximately 53 keV, within the available monochromatic reconstruction range, thus allowing for significant greater detectability. Additional material decomposition technique allows for unique material presentation and analysis such as gadolinium/ water pair analysis with high spatial resolution.

Dual-Energy technology is limited by the types of contrast agents currently available, all based on Iodine. Gadoxetate (Eovist) is a relatively new Gadolinium based MRI contrast agent that is capable of producing not only standard appearing MRI images in the hepatic arterial and portal venous phases, but also provides an opportunity to better visualize the bile ducts and liver parenchyma as it is excreted by the liver into the biliary system during the hepatobiliary phase.

This pilot project aims to address a long-term pitfall in the imaging of cholangiocarcinomas, by providing higher resolution delineation of these often infiltrative tumors on single-source, Dual-Energy Spectral MDCT, capitalizing on improved spatial resolution achievable with MDCT compared to MRI and at the same time producing a non-invasive CT cholangiogram to aid in accurate diagnosis and treatment planning of cholangiocarcinoma, particularly, the hilar variety.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be adult (age 19 or older) with suspected cholangiocarcinoma of the liver.
2. Subject must be able to provide a written informed consent.
3. Subject will be scheduled for gadoxetate contrast enhanced MRI scan of the liver (obtained as part of usual clinical practice).

Exclusion Criteria:

1. Standard MRI safety screening criteria will be employed, and subject will be excluded if any contraindications to undergo MRI are met.
2. Subjects with metallic biliary stents or multiple peripancreatic surgical clips on abdominal MDCT will be excluded.
3. Subjects on hemodialysis or with glomerular filtration rate (GFR) less than 30 will be excluded.
4. Subjects will not be excluded on the basis of gender, race, ethnicity, or religion.
5. Subject may not be pregnant or lactating.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John V Thomas, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gadoxetate Uptake in CT Imaging: Patients will undergo a standard of care Gadoxetate (Eovist 0.025 mmol/kg) MRI for cholangiocarcinoma. Patients will then be immediately placed on the CT scanner. Patients will undergo a dual energy CT of the abdomen with no additional contrast. After the first 8 subjects were accrued, it was apparent that the standard clinical dose was suboptimal for visualization on rsDECT. After obtaining additional regulatory approvals including an investigative New Drug (IND) letter from the FDA, as well as new approval from our institution's IRB, all subsequent subjects were scanned with 0.05 mmol/kg Gadoxetate Disodium. Both groups were injected with Gadoxetate Disodium at a rate of 1 ml/s.
Period: Gadoxetate Standard Dose 0.025 mmol/kg
Arm/Group | Gadoxetate Uptake in CT Imaging
Started | 8
Completed | 8
Not Completed | 0
Period: Gadoxetate Double Dose 0.050 mmol/kg
Arm/Group | Gadoxetate Uptake in CT Imaging
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gadoxetate Uptake in CT Imaging
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [31 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Where Hilar Cholangiocarcinomas Could be Visualized Using Gadoxetate Disodium Enhanced Dual Energy CT
Description: CT scans were assessed for tumor visualization after use of Gadoxetate disodium
Time Frame: 24 hrs
Population: Number of Subjects Where Hilar Cholangiocarcinomas Could be Visualized Using Gadoxetate Disodium Enhanced Dual Energy CT
Measure: Number; unit: participants
Arm/Group | Gadoxetate Uptake in CT Imaging
Number analyzed (Participants) | 18
participants | 5

ADVERSE EVENTS:
Time Frame: Baseline to 24 hours
Arm/Group | Gadoxetate Uptake in CT Imaging
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes